CLINICAL TRIAL: NCT04690114
Title: Incidence, Prevalence. Risk Factors and Epidemiology of SARS-CoV-2 Seropositivity in the Pediatric Population
Brief Title: COVID-10 in the Pediatric Population: SARS-CoV-2 Seropositivity
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shaare Zedek Medical Center (Other)
Collaborators: Ministry of Health, Israel (Other Government)
Responsible Party: Principal Investigator, Adin Breuer, Doctor, Shaare Zedek Medical Center
Other Study IDs: 0387-20-SZMC
Record Dates: First submitted 2020-12-28; First posted 2020-12-30 (Actual); Last update posted 2020-12-31 (Actual); Status verified 2020-12

CONDITIONS: SARS-CoV-2 Infection
Keywords: Serology; SARS-CoV-2 antibodies
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study was to conduct an epidemiological survey of the pediatric population via SARS CoV-2 IgG antibody testing in order to evaluate the incidence of asymptomatic infection and seropositivity among children and establish risk factors of infection and characterization of asymptomatic carriers. Additionally, among seropositive children, antibody titers will be explored in order to reach a better understanding of the relationship between immunity over time after different types of initial exposures.

Methods Study Design and Population A prospective epidemiological survey was conducted in the Pediatric Emergency Department (ED) of the Shaare Zedek Medical Center, a tertiary medical center in Jerusalem, Israel, between October 2020 and January 2021. All patients presenting to the pediatric ED during the study period and requiring blood tests or and IV insertion for any clinical reason were considered eligible to participate in the study. The parents and/or legal guardians of these patients gave oral consent for an additional 1-3 ml of blood to be sent for Sars-CoV-2 antibody testing. In addition, all consenting parent/guardians filled out a comprehensive questionnaire regarding demographic background, past medical history, and specific Covid-19 details such as exposures to carriers, past PCR testing, symptoms etc. All patients with positive serology results were contacted by phone and updated of the test results.

Laboratory testing All blood samples were collected in a clot-activator test tube. Initial testing was conducted using the Abbott SARS-CoV-2 IgG assay. A positive result was considered a value above 1.5 with 0.8 - 1.4 cosidered grayzone results. All positive and grayzone results were then retested in the DiaSoren LIAISON® SARS-CoV-2 S1/S2 IgG assay.

Statistical Analysis Statistical analysis was conducted using SPSS Statistics for Windows, Version 25.0. Armonk, NY: IBM Corp. Clinical variables were analyzed using the Chi-squared test for categorical variables and the t-test for continuous variables. All statistical tests were two-way tests and P value of 5% or less was considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* All patients presenting to the Pediatric Emergency Department for any reason

Exclusion Criteria:

* None

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: All patients presenting to the pediatric ED during the study period and requiring blood tests or and IV insertion for any clinical reason were considered eligible to participate in the study. The parents and/or legal guardians of these patients gave oral consent for an additional 1-3 ml of blood to be sent for Sars-CoV-2 antibody testing. In addition, all consenting parent/guardians filled out a comprehensive questionnaire regarding demographic background, past medical history, and specific Covid-19 details such as exposures to carriers, past PCR testing, symptoms etc. All patients with positive serology results were contacted by phone and updated of the test results.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2020-10-01 (Actual); Primary Completion 2021-05-31 (Estimated); Study Completion 2021-07-31 (Estimated)

PRIMARY OUTCOMES:
Sars-CoV-2 Seropositivity | Six months
  Antibody titers of Sars-CoV-2 antibodies

CONTACTS AND LOCATIONS:
Overall Officials: Eyal Heiman, MD, Principal Investigator — Shaare Zedek Medical Center
Locations (1):
- Shaare Zedek Medical Center, Jerusalem, Israel